CLINICAL TRIAL: NCT00146770
Title: A Multicenter, Multinational, Open-Label Extension Study of the Safety and Efficacy of Aldurazyme® (Laronidase) in Patients With Mucopolysaccharidosis I
Brief Title: Phase 3 Extension Study of the Safety and Efficacy of Aldurazyme® (Laronidase) in Mucopolysaccharidosis I (MPS I) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALID-006-01
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Mucopolysaccharidosis I; Hurler's Syndrome; Hurler-Scheie Syndrome; Scheie Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

ARMS (2):
- Placebo/Aldurazyme (Active Comparator): Patients received placebo for 26 weeks in the Double-Blind Study then received 182 weeks of Aldurazyme (0.58 mg/kg every week) in this Extension Study; patients received a total of 182 weeks of Aldurazyme.
  Interventions: Biological: Aldurazyme; Biological: placebo
- Aldurazyme/Aldurazyme (Active Comparator): Patients received 26 weeks of Aldurazyme in the Double-Blind Study and then received 182 weeks of Aldurazyme in this Extension Study; patients received a total of 208 weeks of Aldurazyme.
  Interventions: Biological: Aldurazyme

INTERVENTIONS:
Biological: Aldurazyme — Placebo for 26 weeks then 0.58 mg/kg Aldurazyme every week for 182 weeks
  Arms: Placebo/Aldurazyme
Biological: Aldurazyme — 0.58 mg/kg Aldurazyme every week for 208 weeks
  Arms: Aldurazyme/Aldurazyme
Biological: placebo — Placebo for 26 weeks
  Arms: Placebo/Aldurazyme

SUMMARY:
This study is being conducted to collect additional long-term efficacy and safety data of Aldurazyme® (laronidase) patients with MPS I disease. Patients who were previously enrolled in the Phase 3 Double-Blind Study will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* The patient or patient's legal guardian must provide written informed consent prior to any protocol-related procedures being performed.
* The patient must have successfully completed Study ALID-003-99 (who received 21 of 26 consecutive weekly infusions).
* The patient has not experienced any safety issues that would contraindicate participation in the Extension study.
* A female patient of childbearing potential must have a negative pregnancy test at entry

Exclusion Criteria:

* The patient is pregnant or lactating.
* The patient has received an investigational drug within 30 days prior to the study enrollment.
* The patient has a medical condition, serious intercurrent illness, or other extenuating circumstance that may significantly interfere with study compliance including all prescribed evaluations and follow-up activities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (25):
- United States (8):
  - University of South Alabama, Mobile, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Toledo Children's Hospital, Toledo, Ohio
  - Merle West Medical Center, Klamath Falls, Oregon
  - The Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
- Brazil (2):
  - Hospital Universatario de Universidade Federal de Santa Catarina, Florianópolis
  - Hospital Infantil Joana de Gusmao, Florianópolis
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Alberta Children's Hospital, Calgary
- Germany (4):
  - Children's Hospital Klinikum Nord Heidberg, Hamburg
  - Medizinishe Hochshule Hannover, Hanover
  - Children's Hospital at the University Hospital of Heidelberg, Heidelberg
  - Children's Hospital Klinikum der F.S. Universitat, Jena
- Catholic University Sacro Cuore, Rome, Italy
- Academisch Ziekenhuis Rotterdam, Rotterdam, Netherlands
- United Kingdom (7):
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Belfast City Hospital, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children and Frenchay Hospital, Bristol
  - Gartnavel Hospital, Glasgow
  - Great Ormond Street Hospital for Sick Children and NHS Trust, London
  - Royal Victoria Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971
- [Derived] Clarke LA, Wraith JE, Beck M, Kolodny EH, Pastores GM, Muenzer J, Rapoport DM, Berger KI, Sidman M, Kakkis ED, Cox GF. Long-term efficacy and safety of laronidase in the treatment of mucopolysaccharidosis I. Pediatrics. 2009 Jan;123(1):229-40. doi: 10.1542/peds.2007-3847. PMID 19117887

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Aldurazyme: Patients received placebo for 26 weeks in the Double-Blind Study then received 182 weeks of Aldurazyme treatment in the Extension Study; patients received a total of 182 weeks of Aldurazyme treatment. "Baseline" for this group is the last measurement in the Double-Bind Study prior to enrollment in this Extension Study.
- Aldurazyme/Aldurazyme: Patients received 26 weeks of Aldurazyme treatment in the Double-Blind Study and then received 182 weeks of Aldurazyme treatment in the Extension Study; patients received a total of 208 weeks of Aldurazyme treatment. "Baseline" for this group is the last measurement prior to randomization in the Double-Blind Study.
Period: Overall Study
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Started | 23 | 22
Completed | 18 | 22
Not Completed | 5 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Aldurazyme: Patients received placebo for 26 weeks in the Double-Blind Study then received 182 weeks of Aldurazyme treatment in the Extension Study; patients received a total of 182 weeks of Aldurazyme treatment.
- Aldurazyme/Aldurazyme: Patients received 26 weeks of Aldurazyme treatment in the Double-Blind Study and then received 182 weeks of Aldurazyme treatment in the Extension Study; patients received a total of 208 weeks of Aldurazyme treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Customized [Number; unit: participants]
  <=12 years | 10 | 12 | 22
  13 to <= 18 years | 8 | 3 | 11
  19 to <= 65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Age characteristics presented were recorded at Baseline in the Double-Blind Study.
  years | 15.4 (7.63) | 15.6 (8.63) | 15.5 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender characteristics presented were recorded at Baseline in the Double-Blind Study.
  Participants
    Female | 12 | 11 | 23
    Male | 11 | 11 | 22
Race/Ethnicity [Number; unit: participants] — Race characteristics presented were recorded at Baseline in the Double-Blind Study.
  participants
    Caucasian | 21 | 16 | 37
    Black | 0 | 0 | 0
    Hispanic | 0 | 4 | 4
    Asian | 1 | 1 | 2
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 182 in Percent Predicted Forced Vital Capacity (FVC)
Description: Percent Predicted Forced Vital Capacity: the maximal exhaled breath volume following a maximal inhaled breath. Overall change from Baseline to Week 182 in percent predicted FVC = (observed value)/(predicted value) * 100%). A higher value indicates a greater response.
Time Frame: Baseline to Week 182
Population: This study enrolled patients who completed the Phase 3 Double-Blind Study and wished to receive open-label treatment with Aldurazyme. The analysis method was intention to treat with last value carried forward.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 23 | 22
percent predicted FVC
  Baseline percentage points FVC | 51.0 (13.15) | 48.4 (14.85)
  Week 182 percentage points FVC | 47.7 (13.69) | 47.2 (15.24)
  Overall Change from Baseline to Week 182 | -3.3 (9.07) | -1.2 (6.52)

2. Primary Outcome: Change From Baseline to Week 182 in Six Minute Walk Test (6MWT)
Description: Six Minute Walk Test: Distance walked (measured in Meters) in 6 minutes. A longer distance indicates a greater response.
Time Frame: Baseline to Week 182
Population: The study enrolled patients who completed the Phase 3 double-blind study and wished to receive open-label treatment with Aldurazyme. The analysis method was intention to treat with last value carried forward.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 23 | 22
Meters
  Baseline distance walked | 348.3 (128.81) | 319.0 (131.41)
  Week 182 distance walked | 367.7 (151.25) | 358.3 (126.40)
  Overall Change from Baseline to Week 182 | 19.4 (107.36) | 39.2 (85.84)

3. Secondary Outcome: Change From Baseline to Week 182 in Apnea/Hypopnea Index (AHI)
Description: Apnea/Hypopnea Index (AHI): Number of absent (apnea) and shallow (hypopnea) breaths per hour of sleep. A greater decrease in events indicates a greater response.
Time Frame: Baseline to Week 182
Population: The study enrolled patients who completed the Phase 3 double-blind study and wished to receive open-label treatment with Aldurazyme. The analysis method was intention to treat.
Measure: Mean (Standard Deviation); unit: Events per Hour
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 15 | 17
Events per Hour
  Baseline events per hour | 14.6 (12.90) | 18.0 (15.54)
  Week 182 events per hour | 9.8 (14.60) | 14.0 (19.32)
  Overall Change from Baseline to Week 182 | -4.8 (13.86) | -4.0 (12.91)

4. Secondary Outcome: Change From Baseline to Week 182 in Liver Volume
Description: Liver Organ Volume: Volume of liver measured by Magnetic Resonance Imaging (MRI). Greater decrease in volume indicates a greater response.
Time Frame: Baseline to Week 182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cubic centimeters (cm3)
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 17 | 21
Cubic centimeters (cm3)
  Baseline liver volume (cm3) | 1351.6 (323.71) | 1228.5 (279.62)
  Week 182 liver volume (cm3) | 1079.9 (256.99) | 1001.4 (157.23)
  Percent Change from Baseline to Week 182 (%) | -17.6 (20.21) | -16.1 (14.76)

5. Secondary Outcome: Change From Baseline to Week 182 in Child Health Assessment Questionnaire/Health Assessment Questionnaire (CHAQ/HAQ) Disability Index Score
Description: CHAQ/HAQ = Patient questionnaire that measures the degree of disability on a scale of 0 (no disability) to 3 (maximal disability). A lower score indicates a greater response.
Time Frame: Baseline to Week 182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 19 | 20
Units on a scale
  Baseline Score | 1.75 (0.740) | 1.99 (0.496)
  Week 182 Score | 1.49 (0.768) | 1.56 (0.758)
  Overall change from Baseline to Week 182 | -0.26 (0.688) | -0.43 (0.574)

6. Secondary Outcome: Change From Baseline to Week 182 in Active Joint Range of Motion (ROM)
Description: Active Joint Range of Motion (ROM): Shoulder Flexion Ability to maximally raise one's arm overhead without assistance. Shoulder range of motion (mean of left and right arms) measured in degrees (0-180) by goniometry. Greater degree of flexion indicates greater response.
Time Frame: Baseline to Week182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 23 | 19
Degrees
  Baseline degrees | 85.2 (32.66) | 96.1 (30.25)
  Week 182 degrees | 103.5 (23.34) | 109.2 (22.24)
  Overall change from Baseline to Week 182 | 18.3 (21.59) | 13.1 (20.66)

7. Other Pre Specified Outcome: Change From Baseline to Week 182 in Urinary GAG Level
Description: Urinary Glycosaminoglycan (GAG) Levels: >> Concentration of GAG relative to creatinine in urine. A greater decrease in GAG level indicates a greater response.
Time Frame: Baseline to Week 182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug GAG/mg Creatinine
Arm/Group | Placebo/Aldurazyme | Aldurazyme/Aldurazyme
Number analyzed (Participants) | 23 | 22
ug GAG/mg Creatinine
  Baseline level (ug GAG/mg Creatinine) | 250.2 (105.09) | 190.2 (59.81)
  Week 182 level (ug GAG/mg Creatinine) | 55.3 (30.88) | 59.8 (34.99)
  Percent change from Baseline to Week 182 (%) | -77.0 (10.09) | -66.3 (21.29)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Placebo/|Aldurazyme***Check Title***: Placebo/|Aldurazyme***Check Description***
- Aldurazyme/|Aldurazyme***Check Title***: Aldurazyme/|Aldurazyme***Check Description***
Arm/Group | Placebo/|Aldurazyme***Check Title*** | Aldurazyme/|Aldurazyme***Check Title***
Serious Adverse Events (participants affected / at risk) | 11/23 | 14/22
Other Adverse Events (participants affected / at risk) | 23/23 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/|Aldurazyme***Check Title*** (N=23) | Aldurazyme/|Aldurazyme***Check Title*** (N=22)
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 | 0
Talipes (Congenital, familial and genetic disorders) | 1 | 0
Corneal opacity (Eye disorders) | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Catheter related complication (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Hernia pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Heart transplant rejection (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Electroencephalogram abnormal (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2
Extensor plantar response (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1
Catheterisation venous (Surgical and medical procedures) | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/|Aldurazyme***Check Title*** (N=23) | Aldurazyme/|Aldurazyme***Check Title*** (N=22)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 2
Splenomegaly (Blood and lymphatic system disorders) | 2 | 4
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 3 | 2
Arrhythmia (Cardiac disorders) | 1 | 2
Atrioventricular block first degree (Cardiac disorders) | 2 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 2
Left atrial dilatation (Cardiac disorders) | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Left ventricular hypertrophy (Cardiac disorders) | 2 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2
Pericardial disease (Cardiac disorders) | 2 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 1
Talipes (Congenital, familial and genetic disorders) | 3 | 2
Cerumen impaction (Ear and labyrinth disorders) | 3 | 2
Deafness (Ear and labyrinth disorders) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 2
Ear disorder (Ear and labyrinth disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 7 | 11
Ear pruritus (Ear and labyrinth disorders) | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 1
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 2
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 4 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 1
Tympanic membrane scarring (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2
Cushingoid (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0
Anisometropia (Eye disorders) | 1 | 0
Astigmatism (Eye disorders) | 1 | 1
Blepharospasm (Eye disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 3
Corneal oedema (Eye disorders) | 1 | 0
Corneal opacity (Eye disorders) | 2 | 5
Dry eye (Eye disorders) | 0 | 1
Eye allergy (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 1 | 2
Eye movement disorder (Eye disorders) | 0 | 1
Eye oedema (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 2 | 2
Eye pruritus (Eye disorders) | 2 | 1
Eye swelling (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Hypermetropia (Eye disorders) | 1 | 1
Hypoaesthesia eye (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 2 | 4
Myodesopsia (Eye disorders) | 1 | 0
Myopia (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1
Papilloedema (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Pseudopapilloedema (Eye disorders) | 0 | 1
Pterygium (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 1 | 1
Retinal pigment epitheliopathy (Eye disorders) | 2 | 1
Strabismus (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 3 | 1
Visual acuity reduced (Eye disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 7 | 9
Abdominal pain lower (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 7 | 8
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 5
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 10
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival cyst (Gastrointestinal disorders) | 1 | 1
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Lip blister (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 12
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 2 | 0
Teething (Gastrointestinal disorders) | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 2 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 6 | 2
Umbilical hernia (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 13 | 12
Application site erythema (General disorders) | 1 | 0
Application site pruritus (General disorders) | 0 | 1
Application site rash (General disorders) | 0 | 1
Asthenia (General disorders) | 2 | 1
Catheter related complication (General disorders) | 2 | 0
Catheter site discharge (General disorders) | 1 | 0
Catheter site erythema (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 2 | 1
Catheter site pain (General disorders) | 3 | 3
Catheter site pruritus (General disorders) | 1 | 1
Catheter site rash (General disorders) | 0 | 2
Catheter site related reaction (General disorders) | 4 | 1
Catheter site swelling (General disorders) | 0 | 1
Catheter site urticaria (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 2
Chest pain (General disorders) | 6 | 7
Chills (General disorders) | 2 | 2
Cyst (General disorders) | 1 | 2
Fatigue (General disorders) | 6 | 9
Feeling cold (General disorders) | 2 | 1
Feeling hot (General disorders) | 3 | 3
Feeling of body temperature change (General disorders) | 2 | 0
Gait disturbance (General disorders) | 6 | 3
Granuloma (General disorders) | 0 | 1
Hangover (General disorders) | 1 | 0
Hernia pain (General disorders) | 1 | 2
Hyperthermia (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 2
Influenza like illness (General disorders) | 3 | 5
Infusion site erythema (General disorders) | 2 | 1
Infusion site extravasation (General disorders) | 4 | 4
Infusion site pain (General disorders) | 3 | 2
Infusion site reaction (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 1
Irritability (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 2 | 4
Pain (General disorders) | 3 | 4
Pyrexia (General disorders) | 16 | 18
Secretion discharge (General disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 5 | 8
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Corneal graft rejection (Immune system disorders) | 2 | 1
Food allergy (Immune system disorders) | 1 | 0
Multiple allergies (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 3
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Central line infection (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 0
Dacryocystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 10 | 7
Enterobiasis (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 1
Herpangina (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 3 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 6 | 1
Laryngitis (Infections and infestations) | 1 | 0
Lice infestation (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 4
Lymph gland infection (Infections and infestations) | 1 | 0
Myringitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 19 | 17
Oral herpes (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 5 | 3
Otitis media (Infections and infestations) | 5 | 6
Otitis media acute (Infections and infestations) | 0 | 2
Otitis media chronic (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 2
Pharyngitis streptococcal (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 3
Postoperative wound infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 4 | 6
Sialoadenitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 4 | 2
Skin infection (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 2 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 7
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 3
Viral diarrhoea (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 2
Viral pharyngitis (Infections and infestations) | 0 | 1
Viral skin infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 5
Device migration (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 3
Extrusion of device (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 3
Incision site pain (Injury, poisoning and procedural complications) | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 7 | 9
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 2
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vena cava injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Bacteria urine (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood iron decreased (Investigations) | 4 | 0
Blood pressure decreased (Investigations) | 0 | 2
Blood pressure diastolic decreased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 4 | 4
Breath sounds abnormal (Investigations) | 0 | 2
Cardiac murmur (Investigations) | 5 | 8
Electrocardiogram PR prolongation (Investigations) | 3 | 1
Electrocardiogram QRS complex abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 3
Eosinophil count increased (Investigations) | 0 | 1
Fungus stool identified (Investigations) | 0 | 1
Grip strength decreased (Investigations) | 1 | 0
Heart sounds abnormal (Investigations) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Mean cell haemoglobin decreased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 2
Renal function test abnormal (Investigations) | 1 | 0
Respiratory rate increased (Investigations) | 1 | 0
Tandem gait test abnormal (Investigations) | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 1
Urine leukocyte esterase positive (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 3 | 1
White blood cells urine positive (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 13
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 4 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint lock (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 4
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 7
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 14
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Unequal limb length (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Aphonia (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 3 | 3
Cervical cord compression (Nervous system disorders) | 0 | 1
Cervical root pain (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 1 | 2
Clumsiness (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2
Coordination abnormal (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 9 | 5
Dizziness postural (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 19 | 19
Hoffmann's sign (Nervous system disorders) | 0 | 2
Hyperreflexia (Nervous system disorders) | 4 | 6
Hypertonia (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 4
Hyporeflexia (Nervous system disorders) | 0 | 2
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Irregular sleep phase (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 3 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0
Loss of proprioception (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 3 | 3
Myoclonus (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 4
Poor quality sleep (Nervous system disorders) | 0 | 1
Post-traumatic headache (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Reflexes abnormal (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 2 | 1
Sensory loss (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 3 | 2
Speech disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Apathy (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Daydreaming (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 4
Disorientation (Psychiatric disorders) | 0 | 1
Flat affect (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 5
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 2
Bilirubinuria (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 2
Enuresis (Renal and urinary disorders) | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 5 | 3
Genital discharge (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Menstrual discomfort (Reproductive system and breast disorders) | 2 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper airway resistance syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 1
Acrodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 3
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Tooth extraction (Surgical and medical procedures) | 2 | 2
Tooth repair (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 3 | 5
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Poor venous access (Vascular disorders) | 4 | 2
Vein disorder (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Rare disease with limited sample size, lack of control group.FVC calculations less reliable for patients whose height is below the 3rdpercent of general population.Height term used to calculate FVC may be influenced by joint contractures and posture.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.